CLINICAL TRIAL: NCT04099095
Title: PROSPECT: A Mental Health Social Prescribing Trial (British Red Cross)
Brief Title: A Mental Health Social Prescribing Trial (British Red Cross)
Acronym: PROSPECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID epidemic
Sponsor: University of South Wales (Other)
Collaborators: British Red Cross (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS 261969
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Mental Health Wellness 1
Keywords: Wait-list

STUDY DESIGN:
Intervention Model Description: The study will employ a randomised wait-list trial design with mixed methods using a co-productive participatory approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Appointment (Active Comparator): Intervention group who receive the Social Prescription without delay. The effectiveness of the consultation and referral process will be assessed
  Interventions: Behavioral: Immediate Appointment
- Delayed Appointment (Active Comparator): Wait-list control group who receive Social Prescribing after a delay of 20 working days. The effectiveness of the consultation and referral process will be assessed
  Interventions: Behavioral: Delayed Appointment

INTERVENTIONS:
Behavioral: Immediate Appointment — The participant will meet the British Red Cross link worker and decide upon a course of action requiring the use of local services appropriate for the participant
  Arms: Immediate Appointment
Behavioral: Delayed Appointment — After a period of delay (control) the participant will meet the British Red Cross link worker and decide upon a course of action requiring the use of local services appropriate for the participant
  Arms: Delayed Appointment

SUMMARY:
Social prescribing is a way of understanding the things that are important to a person and then using these to find groups and resources in their local community that can help them meet their goals and understand their problems. Social prescribing can be used with people who have physical health problems, mental health problems, social problems such as loneliness or financial/housing problems.

The Welsh Government has supported the creation of these social prescribing services across Wales. However, the evidence showing that social prescribing is a good way of improving a person's well-being and quality of life is not very strong.

This project is an evaluation of a new social prescribing service delivered by British Red Cross in two areas in Wales. British Red Cross have made a new social prescribing service, where a link worker works with a patient who has mild/moderate mental or emotional health problems, to understand their needs and set them goals for the future over 12 weeks of core support. The link worker will also help them find services in their local community that might help them achieve their goals.

The study uses a waitlist trial, thus some participants will get to meet the link worker and have the intervention straight away, while others will have to wait for 20 working days. From this, the researchers can compare the people who had the intervention straight away with the people who had to wait. Scores on well-being and quality of life questionnaires will be used to see the effects of the intervention on participants.

DETAILED DESCRIPTION:
Social prescribing is an umbrella term to describe ways of linking people to sources of community-based, non-medical support. There is no fixed definition of social prescribing.

In Wales, social prescribing has many models which require the NHS and third sector organisations to work closely together. These involve referral to a link worker/community connector/social prescriber from primary care or another referral route, such as social work or housing. These roles all practice social prescribing, which includes a 'what matters' conversation, co-productive goal setting, motivational interviewing and coaching, followed by referral to third sector and community groups/professionals for support and activity to meet the person's individual goals.

Social prescribing is being widely implemented and has support from Welsh Government. However, there is limited research evidence to judge its effectiveness, who benefits (if at all) and its value for money. Public Health Wales identified gaps in the published evidence for social prescribing, particularly in the evaluation of social prescribing projects in primary care in Wales. It is therefore important to employ more rigorous and high-quality methods to evaluating social prescribing interventions in the community.

As part of a Welsh Government Third Sector grant for delivering a social prescribing pilot with a focus on mental health, British Red Cross are undertaking a research project in two localities in Wales, Caerphilly and Pembrokeshire, to create and test a model of social prescribing. As part of this initiative, a link worker will work with the individual over a 12-week period to discuss their needs, goals and future steps. A link worker helps the individual to explore extra services that may support them in improving their health, sense of wellness and independence by providing practical and emotional support.

This study will conduct an evaluation alongside the implementation and delivery of the British Red Cross social prescribing intervention, using a randomised waitlist evaluation method. Participants will either receive the social prescribing intervention within 5 days of giving consent, or 20 working days after consent and baseline data collection. This will allow the researchers to draw comparisons between the immediate intervention group and the waitlist controls, who continue to receive usual care. This will also provide a more robust evidence base for social prescribing interventions. The study will use measures of quality of life and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Primary care service users who are at the point of referral
* Experiencing mild/moderate mental health and/or emotional wellbeing disorders( eg anxiety or depression)
* Aged 18+ years
* Registered with a General Practitioner in Wales

Exclusion Criteria:

* Unable to give written informed consent
* Unable to answer all questions (WEMWBS) at baseline
* Worsening of mental health condition to the point where more intensive support is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from base-line. The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) Score | At Base-line, 4 weeks and 3 months after randomisation
  SWEMWBS is completed by the participants and allows self-reflection on mental well-being before and during involvement in health enhancing activities. Each of the 7 statement can be scored from 1 to 5, from 'none of the time' to 'all of the time'. A total score is calculated by summing the 7 individual statement scores. The minimum score is 7 and the maximum is 35. The higher score signifies better mental well-being.
Change from base-line. EQ-5D-5L Health Questionnaire | At Base-line, 4 weeks and 3 months after randomisation
  The EQ-5D-5L Health questionnaire records the self-reported health using five sections: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each section receives a score ranging from 1 to 5, with a score of 5 providing the most ill-health. The minimum total score is 5 and the maximum 25. The lower the score the better the health of the participant. Part 2 of the questionnaire provides a self-reporting vertical visual analogue scale with the end points labelled, "The best health you can imagine" scoring 100 and "The worst health you can imagine", scoring 0.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Llewellyn, Study Director — University of South Wales
Locations (1):
- University of South Wales, Pontypridd, United Kingdom